CLINICAL TRIAL: NCT02643719
Title: Evaluation of a Behavioral Program for Migraineurs in the Emergency Department.
Brief Title: Migraine Treatment in ED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team missed continuing review and study lapsed with out recruiting any subjects.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-01981
Record Dates: First submitted 2015-12-29; First posted 2015-12-31 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Migraine
Keywords: migraine; topiramate
MeSH Terms: conditions — Migraine Disorders | interventions — Relaxation Therapy; Topiramate; Standard of Care; Naproxen; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Topiramate (Active Comparator)
  Interventions: Drug: Topiramate; Drug: Abortive Medication (Naproxen and Sumatriptan)
- Behavioral intervention (Active Comparator)
  Interventions: Behavioral: Relaxation Therapy; Drug: Abortive Medication (Naproxen and Sumatriptan)
- topiramate and behavioral intervention (Active Comparator)
  Interventions: Behavioral: Relaxation Therapy; Drug: Topiramate; Drug: Abortive Medication (Naproxen and Sumatriptan)
- Standard of Care (Active Comparator)
  Interventions: Drug: Standard of Care; Drug: Abortive Medication (Naproxen and Sumatriptan)

INTERVENTIONS:
Behavioral: Relaxation Therapy — Between 30-60 minutes after the standard of care medication administration (metoclopramide, magnesium, prochlorperazine, ketorolac, or steroids at discretion of treating physician), patient receives training in relaxation therapy.
  Arms: Behavioral intervention; topiramate and behavioral intervention
Drug: Topiramate — Preventive medication prescriptions given to the patient along with written instructions and information about side effects:
  Topiramate 25mg tabs (with a plan to increase to 100mg)
  Arms: Topiramate; topiramate and behavioral intervention
Drug: Standard of Care — Standard discharge instruction sheet plus standard of care medication as prescribed by treating physician. The clinical team will be instructed to address post-discharge care as appropriate
  Arms: Standard of Care
Drug: Abortive Medication (Naproxen and Sumatriptan) — All participants will receive abortive medication for acute treatment of their migraine. Preferred medications are Naproxen (500mg) and Sumatriptan (100mg)

SUMMARY:
Randomized pilot feasibility study evaluating the impact of introducing behavioral treatment for migraine in the Emergency Department (ED) and prescribing migraine preventive medications in the ED. The study will examine the effect of these treatments, both individually and in combination, on pain severity and headache-related disability. This study is designed to examine the feasibility of comparing four interventions for ED patients presenting with migraine. Group 1: Starting topiramate; Group 2: Doing a brief behavioral intervention; Group 3: Treating with combination therapy of topiramate and behavioral intervention; and Group 4: Standard of Care.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years to 65 years of age
* primary diagnosis of migraine based on the International Classification of headache disorders 3 beta criteria
* having a migraine 3 or more days/month.

Exclusion Criteria:

* Cognitive Behavioral Therapy (CBT), biofeedback or other relaxation therapy in the past year
* being on medication used for migraine prevention (topiramate, propranolol, valproic acid, amitriptyline/nortriptyline/imipramine/desipramine, botulinum toxin, a SNRI, angiotensin-converting enzyme inhibitors (ACE-I) or ARB)
* cognitive deficit or other physical problem with the potential to interfere with behavioral therapy
* substance or alcohol abuse as determined by self-report or prior documentation in the medical record.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Verbal numeric rating scale (VNRS) scores | 24 hours, 72 hours
  To examine whether there is a significant pain reduction for patients in the ED after behavioral therapy, investigators will analyze pain scores in the ED, and at 24 hours and 72 hours.
Headache Impact Test (HIT) scores | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mia Minen, Principal Investigator — New York University Medical School